CLINICAL TRIAL: NCT05623683
Title: Pain Profiles and Patterns of Physical Activity in Persons With Chronic Knee Pain
Brief Title: P4ACE Trial for Persons With Chronic Knee Pain
Acronym: P4ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: N-20220047
Record Dates: First submitted 2022-11-12; First posted 2022-11-21 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, single-blinded trial, with a 2-arm crossover design.
Who Masked: Participant
Masking Description: To blind the participants, they will be told that both walking interventions are equally likely to cause a decrease, no change, or an increase in knee pain, and we will compare potential differences between the two walking interventions.
  To blind the outcome assessor, the assessor will assess outcomes in a different place from the place where the intervention takes place.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Walking (Active Comparator): Intermittent walking on the treadmill
  Interventions: Other: Intermittent Walking
- Continuous Walking (Active Comparator): Continuous walking on the treadmill
  Interventions: Other: Continuous Walking

INTERVENTIONS:
Other: Intermittent Walking — Wearing comfortable clothes and their usual walking shoes, participants will walk on a treadmill to accrue 30 minutes of walking. Participants will be instructed not to use the treadmill side rails for balance or support during walking. Participants will walk on the treadmill for 3 blocks of 10 minutes with 2 blocks of 5-minute rest (sitting on a chair) in-between. A safety button to stop the treadmill will be available to the participants, so they can stop walking anytime. If participants feel that they are about to lose balance, they are allowed to hold on to the side rails to regain balance and terminate the trial.
  Arms: Intermittent Walking
Other: Continuous Walking — Wearing comfortable clothes and their usual walking shoes, participants will walk on a treadmill to accrue 30 minutes of walking. Participants will be instructed not to use the treadmill side rails for balance or support during walking. Participants will rest for 10 minutes (sitting in a chair) before walking on the treadmill for 1 continuous block of 30 minutes. A safety button to stop the treadmill will be available to the participants, so they can stop walking anytime. If participants feel that they are about to lose balance, they are allowed to hold on to the side rails to regain balance and terminate the trial.
  Arms: Continuous Walking

SUMMARY:
The goal of this single-blind, cross-over clinical trial is to compare the immediate effect of intermittent vs. continuous walking on clinical and mechanistic pain profiles in persons with knee osteoarthritis (OA). In this cross-over trial, participants will perform two types of walking on a treadmill. Intermittent walking will involve 3 blocks of 10 minutes with 2 blocks of 5-minute rest (sitting on a chair) in-between. Continuous walking will involve resting for 10 minutes (sitting in a chair) before walking on the treadmill for 1 continuous block of 30 minutes.

DETAILED DESCRIPTION:
The study objectives are to compare the immediate effect of intermittent vs. continuous walking on clinical and mechanistic pain profiles in persons with knee osteoarthritis (OA). The investigators hypothesize that continuous walking will result in greater increases in clinical pain and mechanistic pain sensitivity than intermittent walking. Physical activity (PA) has been recommended as the first-line management strategy for people with chronic knee pain. Walking is an accessible, low-cost, joint-friendly form of PA and is widely advocated for older adults with knee complaints. However, movement-evoked pain is a commonly cited barrier for PA engagement. On one hand, a bout of PA may produce short-term analgesia and reduce pain. On the other hand, excessive or prolonged PA may exacerbate symptoms and lead to avoidance/fear of subsequent PA. Besides the total PA volume, how it is accumulated could also impact joint health. It is biomechanically plausible that shorter and frequent activities are more beneficial to articular tissues than longer and infrequent activities. Compared to intermittent loading, prolonged continuous loading had a detrimental effect on the biomechanical functions of articular cartilage in a bovine model. Findings of this study will provide insight on the relations between patterns of PA and pain profiles.

ELIGIBILITY:
Inclusion Criteria:

* men or women aged 45-75 years
* BMI ≤ 35 kg/m2
* frequent movement-related knee pain (knee pain on more than half the days of the past month)
* no morning stiffness or morning stiffness lasting < 30-min
* self-reported unilateral or bilateral knee pain of ≥ 3 and ≤ 7 on a 0-10 numeric pain rating scale (NPRS)
* knee pain duration ≥ 12 months
* physically able to walk unassisted on a treadmill at ≥ 4 km/hour for 30 minutes
* own a smart phone
* willing and able to wear an activity monitor and answer electronic survey questions delivered via a smart phone over a 10-day period.

Exclusion Criteria:

* intra-articular steroid injections in the previous 3 months
* intra-articular hyaluronic acid injection in the previous 6 months
* any arthroscopic or surgical knee procedures (e.g., partial meniscectomy) in the past 12 months
* lumbar radiculopathy
* neurological, vestibular, or visual dysfunction affecting walking balance and mobility
* plan for total knee arthroplasty in the next 12 months

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change from pre-walking to immediately post-walking in Numeric Pain Rating Scale (NPRS) for current knee pain | pre-walking, immediately post-walking
  The primary outcome is the self-reported clinical pain. The pre- and post-walking knee pain will be rated right before the commencement of the walking program and at the termination of the walking program respectively. Participants verbally select a value that corresponds with the intensity of pain that they experience. "0" means "no pain" and "10" means "pain as bad as you can imagine" or "worst pain imaginable". The NPRS, an 11-point (i.e., 0-10) measure of pain intensity, is recommended as a core outcome measure in clinical trials of chronic pain treatments and has excellent reliability and validity for adults with chronic musculoskeletal pain. On average, a change of 2 points or a change of approximately 30% in NPRS represented a clinically important difference in adults with chronic pain.

SECONDARY OUTCOMES:
Change from pre-walking to immediately post-walking in Cuff Pain Detection Threshold (cPDT) | pre-walking, immediately post-walking
  A computer-controlled cuff algometer will measure cPDT. Participants will be fitted with 13-cm-wide silicone tourniquet cuffs (VBM, Düsseldorf, Germany) on bilateral lower limbs. The cuff inflation will be controlled by a cuff algometry system (Cortex Technology, Hadsund, Denmark). The cuff will be inflated at a rate of 1kPa/s to a maximum of 100 kPa. Using a hand-held electronic device with a release button for deflating the cuff, participants will be instructed to rate the pressure pain continuously on a 10-cm visual analogue scale (VAS), until the pain becomes intolerable, at which point they will press the release button to terminate the test. The cPDT will be the cuff pressure reading at the time of VAS rating of 1cm. The cuff-system is user independent and has been shown to be reliable for the outcomes assessed.
Change from pre-walking to immediately post-walking in Cuff Pain Tolerance Threshold (cPTT) | pre-walking, immediately post-walking
  A computer-controlled cuff algometer will measure cPDT. Participants will be fitted with 13-cm-wide silicone tourniquet cuffs (VBM, Düsseldorf, Germany) on bilateral lower limbs. The cuff inflation will be controlled by a cuff algometry system (Cortex Technology, Hadsund, Denmark). The cuff will be inflated at a rate of 1kPa/s to a maximum of 100 kPa. Using a hand-held electronic device with a release button for deflating the cuff, participants will be instructed to rate the pressure pain continuously on a 10-cm visual analogue scale (VAS), until the pain becomes intolerable, at which point they will press the release button to terminate the test. The cPTT will be the cuff pressure reading at the time of test termination (i.e., when the pain becomes intolerable). If the tolerance threshold is not achieved before the 100 kPa limit, cPTT will be 100 kPa. The cuff-system is user independent and has been shown to be reliable for the outcomes assessed.
Change from pre-walking to immediately post-walking in Temporal Summation of Pain (TSP) | pre-walking, immediately post-walking
  Using the same cuff algometry system, the TSP will be assessed by delivering 10 rapid cuff pressure stimuli at a pressure magnitude of the cPTT lasting for one second. Each stimulus will be followed by 1-second break before the next stimulus. Participants will be instructed to rate the pain intensity on the electronic VAS for each stimulus without returning the VAS to zero between inflations. The VAS score will be recorded for each stimulus. This procedure has been shown to be reliable with Intraclass Correlation Coefficients of 0.70-0.77.
Change from pre-walking to immediately post-walking in Conditioned Pain Modulation (CPM) | pre-walking, immediately post-walking
  The CPM will be assessed by re-measuring the cPDT of the index limb during a simultaneously painful conditioning stimulus on the non-index limb. An increase in cPDT from baseline would indicate a CPM response.

CONTACTS AND LOCATIONS:
Overall Officials: Alison H Chang, Principal Investigator — Aalborg University; Michael Rathleff, Study Director — Aalborg University
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No